CLINICAL TRIAL: NCT04110171
Title: Relationship Between the Nutritional Habits and Relapsing and Disability Rates in Patient With
Brief Title: Relationship Between the Nutritional Habits and Relapsing and Disability Rates in Patient With Multiple Sclerosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Abd alazeem Moustafa, investigator, Assiut University
Other Study IDs: nutritional habits in multiple
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Nutrition Habits in Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
patient with multiple sclerosis will undergo and completed comprehensive survey measuring body mass index and assessment of obesity ,health related quality of life,disability,relapsing and complete data on their dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years of age
* males or females
* all cases of diagnosed multiple sclerosis under treatment or not

Exclusion Criteria:

* disable cases
* long standing disease more than five years.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patient 20 and 40 years ago with both gender diagnosed with multiple sclerosis under treatment or not
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
measurement of the body mass index and so assessment of obesity of the patient and multiple sclerosis . also assessment of nutrition habits by dietary habits questionnaire in theses patient . | one and half year
  dietary habits questionnaire include
  * family eating habits
  * personal dietary assessment personal eating habits
  * personal back ground information The questionnaire considers both the type of food consumed and the methods of food preparation. Each item scores from 1 to 5 with a score of 1 indicating very poor dietary behavior and a score of 5 indicating healthy.These items give rise to 10 dietary sub scores: cereals, fruit and vegetables, omega-3 fatty acids, food choices, food preparation, takeaways and snacks, fat, fiber, sodium, Mean scores ranging from 1 to 5 are calculated for each sub score
assessment of disability rates of the patient of multiple sclerosis. | one and half year
  the disability rate assessed by expanded disability status scale which is a self-reported surrogate tool used by neurologists to assess gait disability.33,34 Th scored ordinally from 0 (normal) to 8 (bed bound).
  bound)